CLINICAL TRIAL: NCT00535301
Title: Outcome After Anterior Vaginal Prolapse Repair: A Randomized Controlled Trial
Brief Title: Outcomes of Anterior Colporrhaphy Versus Graft Reinforced Anterior Prolapse Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4348
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cystocele; Uterine Prolapse; Urinary Incontinence
Keywords: cystocele; uterine prolapse; urinary incontinence
MeSH Terms: conditions — Cystocele; Uterine Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior Colporrhaphy (sutured repair) (Placebo Comparator): Anterior vaginal prolapse repair with anterior colporrhaphy (no graft) using sutures.
  Interventions: Procedure: sutured anterior vaginal prolapse repair
- Perigee (grafted repair) (Active Comparator): Anterior vaginal prolapse repair with graft
  Interventions: Device: grafted anterior prolapse repair

INTERVENTIONS:
Device: grafted anterior prolapse repair — anterior vaginal prolapse repair with graft
  Other Names: Perigee Transobturator Prolapse Repair System
  Arms: Perigee (grafted repair)
Procedure: sutured anterior vaginal prolapse repair — anterior vaginal prolapse repair with suture
  Other Names: cystocele repair
  Arms: Anterior Colporrhaphy (sutured repair)

SUMMARY:
The purpose of this study is determine whether grafted anterior vaginal prolapse repair is more effective and associated with less complications than prolapse repair with suture.

DETAILED DESCRIPTION:
Successful correction of anterior vaginal prolapse remains one of the most challenging aspects of pelvic reconstructive surgery. Up to 70% have recurrent prolapse following anterior colporrhaphy. The low success rate has consequently led to widespread use of grafts in anterior vaginal prolapse repair. While both biologic grafts and polyglactin 910 mesh have yielded disappointing results, uncontrolled studies have demonstrated low recurrence rates with polypropylene mesh reinforcement.

The Perigee Transobturator Prolapse Repair System (Perigee TPRS) (American Medical Systems, Minnetonka, Minnesota) is used to repair anterior vaginal prolapse via a transobturator approach. Specially-designed helical needles are utilized to attach either a porcine dermal (InteXenTM) or soft polypropylene (InteProTM) graft to the pelvic sidewall at four points. We designed this randomized control trial to compare the anatomic success rates, effect on quality of life and sexual symptom scores, and rates of adverse events of the Perigee TPRS with polypropylene mesh to that of anterior colporrhaphy.

ELIGIBILITY:
Inclusion Criteria:

* stage II or greater anterior vaginal prolapse requiring surgical correction
* age 21 years and older

Exclusion Criteria:

* less than Stage II anterior vaginal prolapse
* decline participation
* pregnant or contemplating future pregnancy
* prior anterior vaginal prolapse repair with biologic or synthetic graft
* active or latent systemic infection
* compromised immune system
* previous pelvic irradiation or cancer
* known hypersensitivity to polypropylene
* uncontrolled diabetes mellitus
* unable or unwilling to give valid informed consent
* unable or unwilling to comply with the protocol
* scheduled to undergo concomitant Burch colposuspension or pubovaginal sling

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N Nguyen, MD, Principal Investigator — Southern California Permanente Medical Group
Locations (1):
- Kaiser Permanente, Downey, California, United States

REFERENCES:
- [Background] Gauruder-Burmester A, Koutouzidou P, Rohne J, Gronewold M, Tunn R. Follow-up after polypropylene mesh repair of anterior and posterior compartments in patients with recurrent prolapse. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Sep;18(9):1059-64. doi: 10.1007/s00192-006-0291-7. Epub 2007 Jan 12. PMID 17219252
- [Derived] Nguyen JN, Burchette RJ. Outcome after anterior vaginal prolapse repair: a randomized controlled trial. Obstet Gynecol. 2008 Apr;111(4):891-8. doi: 10.1097/AOG.0b013e31816a2489. PMID 18378748

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Female Pelvic Medicine and Reconstructive Surgery Clinic at Kaiser Permanente Bellflower Medical Center between January 2005 and April 2006.
Pre-assignment Details: Exclusion criteria were less than stage II anterior vaginal prolapse, current or future pregnancy, prior grafted anterior prolapse repair, impaired wound healing, known hypersensitivity to polypropylene, unable or unwilling to give valid informed consent or if scheduled to undergo concomitant Burch colposuspension or pubovaginal sling.
Groups:
- Anterior Colporrhaphy: Anterior vaginal prolapse repair with anterior colporrhaphy (no graft)
- Perigee: Anterior vaginal prolapse repair with graft
Period: Overall Study
Arm/Group | Anterior Colporrhaphy | Perigee
Started | 38 | 38
Completed | 33 | 33
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Colporrhaphy | Perigee | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.5) | 61 (10.5) | 60 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Stage II or Greater Anterior Vaginal Prolapse
Description: Pelvic Organ Prolapse Quantification Point Ba is the most distal position of any part of the anterior vagina between point Aa and the vaginal cuff or anterior vaginal fornix. Better vaginal support is assigned a negative value (ie, if there is no prolapse, point Ba is -3 cm by definition). Vaginal prolapse beyond the hymen, indicating worse vaginal support, is assigned a positive value (this may be equal to the total vaginal length at the maximum). Recurrent stage II or greater anterior vaginal prolapse is defined as POPQ Point Ba measurement equal to or greater (more positive) than -1.
Time Frame: three years
Population: Intention to Treat. Stage II or greater anterior vaginal prolapse was defined as POPQ Ba equal to or greater than -1.
Measure: Number; unit: participants
Arm/Group | Anterior Colporrhaphy | Perigee
Number analyzed (Participants) | 38 | 38
participants | 24 | 11
Statistical Analysis 1: Comparison: Anterior Colporrhaphy vs Perigee; Sample size was calculated based on previously-published anatomic success rates of standard anterior colporrhaphy (50%) and polypropylene mesh-reinforced anterior vaginal repair (85%) (1-10). Assuming a 2-sided hypothesis test with 5% type I error and 80% power, 33 patients in each group would be required to detect an absolute difference of 35% or more in recurrent stage II prolapse. Assuming a 15% drop-out rate, we sought to enroll 76 patients into the clinical trial; Test type: Superiority or Other; p = 0.005, Chi-squared; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.1 to 0.6], Standard Deviation 2

2. Secondary Outcome: Operative Time
Description: Calculated as time from first incision to time of closure of last incision.
Time Frame: perioperative
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Anterior Colporrhaphy (Sutured Repair): Sutured anterior vaginal prolapse repair with anterior colporrhaphy (no graft)
Arm/Group | Anterior Colporrhaphy (Sutured Repair) | Perigee (Grafted Repair)
Number analyzed (Participants) | 38 | 38
minutes | 120 [60 to 150] | 135 [65 to 210]
Statistical Analysis 1: Comparison: Anterior Colporrhaphy (Sutured Repair) vs Perigee (Grafted Repair); Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Vaginal Mesh Exposure
Description: Vaginal mesh exposure defined as appearance of mesh, placed during the index surgery, not covered by overlying vaginal epithelium on postoperative pelvic exams subsequent to the first postoperative exam. May be either symptomatic or asymptomatic. This was not differentiated in the statistical analysis.
Time Frame: perioperative
Measure: Number; unit: participants
Arm/Group | Anterior Colporrhaphy | Perigee
Number analyzed (Participants) | 38 | 38
participants | 0 | 4
Statistical Analysis 1: Comparison: Anterior Colporrhaphy vs Perigee; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: three years
Arm/Group | Anterior Colporrhaphy | Perigee
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/37

LIMITATIONS AND CAVEATS:
-Small number of subjects, Single surgeon, Medium follow-up, Limited ability to detect uncommon adverse events and small differences in quality of life and sexual symptom scores, Concurrent pelvic reconstructive and anti-incontinence procedures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No